CLINICAL TRIAL: NCT04603690
Title: Complementary Therapy of Dietary Supplements Curcumin, Quercetin and Vitamin D3 for Mild to Moderate Symptoms of COVID-19
Brief Title: Oral Curcumin, Quercetin and Vitamin D3 Supplements for Mild to Moderate Symptoms of COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ikram Din Ujjan, MBBS, PhD, Professor of Pathology, Liaquat University of Medical & Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LUMHS/REC/173
Record Dates: First submitted 2020-10-24; First posted 2020-10-27 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19 | interventions — Complementary Therapies; Standard of Care

STUDY DESIGN:
Intervention Model Description: Pilot, randomized, controlled, open-label and pragmatic trial, comparing the treatment benefits of combination of curcumin, quercetin and vitamin D3 supplements as add-on to standard treatment vs. standard therapy, in mild to moderate symptomatic COVID-19 outpatients, within 48 hours, for testing Positive for SARS-CoV-2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Complementary therapy group (Experimental): This arm will receive a daily supplementation of 168 mg curcumin, 260 mg quercetin and 9 mcg/360 IU of vitamin D3 (cholecalciferol) as add-on to the standard of care for 14-days
  Interventions: Dietary Supplement: Complementary therapy; Drug: Standard of care
- Control group (Active Comparator): This arm will receive standard care alone
  Interventions: Drug: Standard of care

INTERVENTIONS:
Dietary Supplement: Complementary therapy — A daily supplementation of 168 mg curcumin, 260 mg quercetin and 360 IU of vitamin D3 (cholecalciferol) for 14-days
  Arms: Complementary therapy group
Drug: Standard of care — This arm will receive standard of care as per the hospital guidelines

SUMMARY:
The present study is aimed to investigate the treatment benefits of a combination of dietary supplements quercetin, curcumin and vitamin D3 as add-on therapy to the routine care for early mild symptoms of COVID-19 infection in outpatients setting.

DETAILED DESCRIPTION:
There is currently no specific early-stage therapeutic treatment available for COVID-19.

Dietary supplements curcumin, quercetin and vitamin D3 have shown strong antioxidant, anti-inflammatory/immunomodulatory and broad-spectrum antiviral effects. The present study is focused to test the combination of oral curcumin, quercetin and vitamin D3 supplements as complementary therapy for outpatients with mild to moderate symptoms of COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older, of either gender
* Patients must be tested positive for SARS-CoV-2 by RT-PCR within 72 hours prior to enrolment
* Patients must exhibit typical symptoms of COVID-19 disease at screening such as fever, fatigue, a dry and contagious cough, loss of appetite, body aches, shortness of breath, mucus or phlegm, sore throat, headache, chills, sometimes with shaking, loss of smell or taste, congestion or runny nose, nausea, or vomiting, diarrhea, muscular pain etc.
* Patients must be in the early stage of COVID-19 disease who do not require hospitalization at the time of screening
* Patients must be under the care of a Physician for diagnosis of COVID-19
* Patients who have signed informed consent

Exclusion Criteria:

* Patients with proven hypersensitivity or allergic reaction to quercetin or curcumin
* Patients with known chronic kidney disease with estimated creatinine clearance < 50 mL/minute or need for dialysis
* Patients who are severely hypotensive defined as needing hemodynamic pressors to maintain blood pressure
* Patients taking anticoagulant/antiplatelet drugs such as Coumarine, Heparine, Aspirin, Clopidrogel, dalteparin, enoxaparin, ticlopidine and warparin.
* Patients with gallstone obstruction
* Hypothyroid suffering patients
* Patients with moderate or severe thrombocytopenia (platelet count <100 ×10⁹/L);
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 Negativity by RT-PCR | up to 14 days
  Number of patients testing negative for COVID-19
COVID-19 symptoms improvement | up to 7 days
  Number of patients with improvement in COVID-19 acute symptoms

SECONDARY OUTCOMES:
Improvement in the serum inflammatory marker level | up to 7 days
  Changes in the serum CRP level
Improvement in the serum inflammatory marker level | up to 7 days
  Changes in the serum D-dimer level
Improvement in the serum inflammatory marker level | up to 7 days
  Changes in the serum LDH level
Improvement in the serum inflammatory marker level | up to 7 days
  Changes in the serum ferritin level
Hospitalization rate | up to 14 days
  Number of patients required hospitalization
Length of hospitalization | up to 14 days
  Number of hospital admission days
Length of supplementary oxygen therapy | up to 14 days
  Patients requirement oxygen at during hospitalization
ICU transfer | up to 14 days
  Numbers of patients progressing to ICU
Mechanical ventilation | up to 14 days
  Numbers of patients requiring mechanical ventilation at hospital
All cause mortality | up to 14 days
  Numbers of hospital mortality
Safety and tolerability | up to 14 days
  Any adverse event due to the investigational treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Liaquat University Hospital, Jāmshoro, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ujjan ID, Khan S, Nigar R, Ahmed H, Ahmad S, Khan A. The possible therapeutic role of curcumin and quercetin in the early-stage of COVID-19-Results from a pragmatic randomized clinical trial. Front Nutr. 2023 Jan 18;9:1023997. doi: 10.3389/fnut.2022.1023997. eCollection 2022. PMID 36742008